CLINICAL TRIAL: NCT07147803
Title: Sleep Quality in Patients With Non-cystic Fibrosis Bronchiectasis in Asyut University Hospitals: Correlation With Clinical, Functional, and Radiological Parameters
Brief Title: Sleep Quality in Patients With Non-cystic Fibrosis Bronchiectasis
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Montaser Gamal Ahmed, Lecturer of Chest Diseases and Tuberculosis, Assiut University
Other Study IDs: MGAhmed-Sleep-Bronchiectasis
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bronchiectasis; Sleep-Disordered Breathing
Keywords: Bronchiectasis; Sleep; Quality of life; Exacerbations
MeSH Terms: conditions — Bronchiectasis; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bronchiectasis Patients: Confirmed non-CF bronchiectasis on high-resolution CT (HRCT) by a chest radiologist, with standard features (e.g., broncho-arterial ratio >1, lack of tapering, airways visible within 1 cm of pleura), documented in the medical record
  Interventions: Other: Pittsburgh Sleep Quality Index

INTERVENTIONS:
Other: Pittsburgh Sleep Quality Index — PSQI (Arabic validated version) - main sleep measure; global score 0-21; PSQI >5 = poor sleep quality.

SUMMARY:
Non-cystic fibrosis (non-CF) bronchiectasis is a chronic, heterogeneous airway disease characterized by irreversible bronchial dilatation, persistent airway infection, and neutrophilic inflammation that together drive daily cough, sputum production, recurrent exacerbations, and progressive functional decline. Sleep is a key determinant of Health-Related Quality of Life (HRQoL) and cardiometabolic health. In chronic lung diseases, nocturnal hypoxemia, cough, dyspnea, and systemic inflammation commonly disrupt sleep continuity and architecture. In bronchiectasis specifically, several studies show high rates of poor sleep quality using the Pittsburgh Sleep Quality Index (PSQI), with ~50-60% of clinically stable patients classified as "poor sleepers," often accompanied by daytime dysfunction. Poor sleep correlates with disease severity indices and symptoms such as nocturnal cough.

DETAILED DESCRIPTION:
In Egypt, bronchiectasis is a frequent clinical problem seen across tertiary hospitals. Recent tertiary-center studies from Upper Egypt (including Asyut) have described the prevalence and early outcomes of bronchiectasis among admitted adults, underscoring its local clinical significance. However, despite multiple Egyptian works on sleep quality in other respiratory conditions (e.g., COPD) using the PSQI, there remains a clear evidence gap regarding sleep quality specifically in adult non-CF bronchiectasis. International cohorts consistently demonstrate prevalent sleep disturbance in bronchiectasis and links to clinical severity, but Egyptian data in non-CF adult bronchiectasis are scarce. Locally contextualized evidence is needed to understand whether sleep impairment in our patients aligns with international observations and how it relates to spirometric function, structural disease burden, composite severity indices, and inflammatory biomarkers within an Upper Egypt setting.

Our study aims to Quantify sleep quality using the PSQI in adults with non-CF bronchiectasis attending Asyut University Hospitals, and Evaluate its correlations with clinical parameters (symptoms, exacerbations, mMRC, Quality of Life)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (adults).
* Confirmed non-CF bronchiectasis on high-resolution CT (HRCT) by a chest radiologist, with standard features (e.g., broncho-arterial ratio >1, lack of tapering, airways visible within 1 cm of pleura), documented in the medical record.
* Non-cystic fibrosis etiology: no clinical diagnosis of cystic fibrosis; if prior doubt, a negative/normal sweat chloride or genetic report will be needed.

Exclusion Criteria:

* Acute exacerbation at screening or within the preceding 4 weeks, or need for systemic antibiotics or systemic corticosteroids in that window.
* Severe hemoptysis, unstable respiratory status, or any condition where completing questionnaires/testing is unsafe per investigator.
* Primary sleep disorders that would cloud PSQI interpretation unless stable ≥3 months (e.g., moderate-severe OSA newly diagnosed and initiating PAP therapy; narcolepsy; untreated restless legs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age ≥18 years (adults).
  * Confirmed non-CF bronchiectasis on high-resolution CT (HRCT) by a chest radiologist, with standard features (e.g., broncho-arterial ratio >1, lack of tapering, airways visible within 1 cm of pleura), documented in the medical record.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of poor sleep | 24 hours
  (PSQI > 5)

CONTACTS AND LOCATIONS:
Overall Officials: Montaser Gamal, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao Y, Guan W, Xu G, Lin Z, Tang Y, Lin Z, Li H, Gao Y, Luo Q, Zhong N, Chen R. Sleep disturbances and health-related quality of life in adults with steady-state bronchiectasis. PLoS One. 2014 Jul 18;9(7):e102970. doi: 10.1371/journal.pone.0102970. eCollection 2014. PMID 25036723
- [Background] Martinez-Garcia MA, Athanazio RA, Giron R, Maiz-Carro L, de la Rosa D, Olveira C, de Gracia J, Vendrell M, Prados-Sanchez C, Gramblicka G, Corso Pereira M, Lundgren FL, Fernandes De Figueiredo M, Arancibia F, Rached SZ. Predicting high risk of exacerbations in bronchiectasis: the E-FACED score. Int J Chron Obstruct Pulmon Dis. 2017 Jan 18;12:275-284. doi: 10.2147/COPD.S121943. eCollection 2017. PMID 28182132